CLINICAL TRIAL: NCT02639286
Title: A Randomized, Double Blind, Placebo-Controlled Study to Assess Efficacy, Safety and Tolerability of ISIS 304801 in Patients With Partial Lipodystrophy With an Open-Label Extension
Brief Title: Efficacy, Safety and Tolerability of ISIS 304801 in People With Partial Lipodystrophy With an Open-Label Extension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 160038; 16-DK-0038 (Other: NIH Clinical Center)
Record Dates: First submitted 2015-12-23; First posted 2015-12-24 (Estimated); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-01-03

CONDITIONS: Lipodystrophy
Keywords: Lipodystrophy; Hypertriglyceridemia
MeSH Terms: conditions — Lipodystrophy; Hypertriglyceridemia | interventions — ISIS 304801

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo administered subcutaneously (SC)
  Interventions: Drug: Placebo
- ISIS 304801 (Experimental): 300 mg of study drug administered via SC
  Interventions: Drug: ISIS 304801

INTERVENTIONS:
Drug: ISIS 304801 — 300 mg of ISIS 304801 administered as SC
  Arms: ISIS 304801
Drug: Placebo — Placebo administered via SC
  Arms: Placebo

SUMMARY:
Background:

Partial lipodystrophy is a deficiency of body fat in parts of the body (usually the arms and legs). People with partial lipodystrophy often get high blood triglyceride (fat) level, insulin resistance, diabetes and other problems. Researchers think the new drug ISIS 304801 can help treat health problems caused by partial lipodystrophy.

Objective:

To see if ISIS 304801 will improve blood fat (triglyceride levels), diabetes, and liver disease, and reduce some risks for heart disease caused by partial lipodystrophy.

Eligibility:

Adults at least 18 years old with partial lipodystrophy.

Design:

Participants will be screened during a 1-week stay at NIH. They will have:

Blood and urine tests

Physical exam.

Assignment to get either the study drug or placebo.

Instructions for how to inject the drug.

Body measurements.

Heart tests.

Participants will give themselves injections of the drug or placebo once a week at home. Some may test blood sugar by finger pricks. They will have monthly phone calls and nurse visits to take blood tests.

After 4 months, participants may continue the study for 1 year. All participants will get the study drug.

Participants will have study visits at NIH every 4 months. These may include:

Insulin sensitivity measurement: Insulin and sugar will be infused through 2 intravenous (IV) lines in the arms. Blood will be drawn.

Sugar and fat metabolism measured by IV infusions and blood tests.

Special x-ray scan to measure body fat.

Liquid meal then blood collected by IV catheter in the arm.

Magnetic resonance imaging scans.

Neck ultrasound.

Questionnaires.

Liver biopsy (optional)

Injection of heparin (a blood thinner) before a blood test.

After finishing the drug, participants will have 1 nurse visit and 1 visit to NIH.

...

DETAILED DESCRIPTION:
Background:

Lipodystrophy is a rare disease of deficient adipose mass, characterized by severe hypertriglyceridemia as well as insulin resistance, diabetes mellitus, fatty liver disease, acute pancreatitis, and early cardiovascular events. Apolipoprotein C-III (apoC-III) regulates triglyceride metabolism, and apoC-III levels strongly correlate with serum triglycerides in a variety of patient populations. Patients with genetically low levels of apoC-III have lower triglycerides and reduced cardiovascular disease, while individuals with genetically elevated levels of apoC-III have higher triglycerides and increased non-alcoholic fatty liver disease and insulin resistance. Pharmacologic reduction of apoC-III using anti-sense oligonucleotides (ASOs) reduce triglycerides by ~60-70% in a tested patient populations.

Aim:

The purpose of this study is to determine if apoC-III reduction using an ASO to apoC-III (ISIS 304801) will reduce triglycerides and improve insulin resistance, diabetes, and hepatic steatosis in patients with lipodystrophy.

The primary hypothesis to be tested is:

1. ISIS 304801will reduce log10 fasting serum triglycerides.

   Secondary and tertiary hypotheses to be tested are:
2. ISIS 304801will improve glucose metabolism by improving insulin resistance.
3. ISIS 304801 will reduce hepatic steatosis.
4. ISIS 304801 will improve cardiovascular risk markers.

We will also explore the mechanism of action of apoC-III ASO by studying lipoprotein lipase activity and lipoprotein particle distribution.

Methods:

This study will enroll up to 20 patients with partial lipodystrophy with a goal of 10 study completers. The study will be conducted in two phases. The first is a 16-week, randomized, double-blind, placebo-controlled design. Subjects will be treated with ISIS 304801 at a target dose of 300 mg per week or placebo. Following this phase, all subjects will enter a 12 month open-label extension in which they will receive active drug. Patients who experience benefit (triglyceride lowering greater than or equal to 50%) may receive an additional 12 months of open-label drug (up to 24 months, total). Measurement of the primary outcome (serum triglycerides) and key secondary outcomes will be performed at baseline prior to the intervention, after 13 weeks (primary outcome only) or 16 weeks (primary and secondary outcomes) of blinded drug or placebo, and after an additional 4 months of active drug in subjects initially randomized to placebo.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18 years at enrollment (the time of informed consent, week -1)
* Fasting triglyceride (TG) levels greater than or equal to 500 mg/dL (greater than or equal to 5.7 mmol/L) at enrollment. If the fasting TG value is <500 mg/dL (<5.7 mmol/L) but greater than or equal to 350 mg/dL (greater than or equal to 4.0 mmol/L) up to two additional tests may be performed in order to qualify, and a single level greater than or equal to 500 mg/dL will permit enrollment.

OR

* Fasting TG levels greater than or equal to 200 mg/DL (2.6 mmol/L) with a hemoglobin A1C over 7%.
* Willing to maintain their customary physical activity level and to follow a diet moderate in carbohydrates and fats with a focus on complex carbohydrates and replacing saturated for unsaturated fats
* Clinical diagnosis of lipodystrophy based on deficiency of subcutaneous body fat in a partial fashion assessed by physical examination, and low skinfold thickness in anterior thigh by caliper measurement: men (less than or equal to 10mm) and women (less than or equal to 22mm), plus one of the following:

  * Genetic diagnosis of familial PL (e.g., mutations in LMNA, PPARG, AKT2, or PLIN1 genes) OR

    * Family history of familial PL or abnormal and similar fat distribution plus 1 minor criterion (below), OR
    * 2 minor criteria (below) in the absence of genetic diagnosis of family history
    * MINOR Criteria
    * Diabetes mellitus with requirement for high doses of insulin, eg, requiring greater than or equal to 200 U/day,greater than or equal to 2 U/kg/day, or currently taking U-500 insulin
    * Presence of acanthosis nigricans on physical examination
    * History of polycystic ovary syndrome (PCOS) or PCOS-like symptoms (hirsutism, oligomenorrhea, and/or polycystic ovaries)
    * History of pancreatitis associated with hypertriglyceridemia
    * Evidence of non-alcoholic fatty liver disease: Hepatomegaly and/or elevated transaminases in the absence of a known cause of liver disease or Radiographic evidence of hepatic steatosis (e.g., on ultrasound or CT)
* Satisfy one of the following:

  * Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females >55 years of age or, in females less than or equal to 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and follicle-stimulating hormone (FSH) levels in the postmenopausal range for the laboratory involved), abstinent, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method from time of signing the informed consent form until at least 13 weeks after the last dose of Study Drug administration.
  * Males: Surgically sterile, abstinent, or if engaged in sexual relations with a female of child bearing potential, patient is utilizing an acceptable contraceptive method from the time of signing the informed consent form until at least 13 weeks after the last dose of study drug administration.

Note: Abstinence is only an effective method of birth control when this is the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception.

EXCLUSION CRITERIA:

* A diagnosis of generalized lipodystrophy
* Current or history of autoimmune diseases (even with a diagnosis of PL) unless approved by the Investigator and Sponsor Medical Monitor
* Acute pancreatitis within 4 weeks of enrollment
* History within 6 months of enrollment of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack, or unstable congestive heart failure requiring a change in medication
* Major surgery within 3 months of enrollment
* History of heart failure with New York Heart Association functional classification (NYHA) greater than Class II
* Uncontrolled hypertension (blood pressure [BP] >160/100 mm Hg)
* Any of the following laboratory values at enrollment:

  * Cardiac troponin T > upper limit of normal (ULN)
  * Measured or estimated (in case of triglycerides > 400 mg/dL) LDL-C >130 mg/dL on maximal tolerated statin therapy
  * Hemoglobin HbA1c greater than or equal to 9.5%
  * Hepatic:

    * Total bilirubin >ULN
    * Alanine transaminase (ALT) >3.0 x ULN. Higher levels will be permitted after a safety review by a hepatologist, that includes no evidence of cirrhosis.
    * Aspartate aminotransferase ( (AST) >3.0 x ULN. Higher levels will be permitted after a safety review by a hepatologist, that includes no evidence of cirrhosis.
  * Renal:

    * Persistently positive (2 out of 3 tests greater than or equal to trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing less than or equal to 5 red blood cells per high power field (urine will be screened at admission and repeated if abnormal). If red blood cell counts (RBC) are high every effort will be made to determine if the source is renal or benign, such as from menstrual bleeding. If the presence of RBC is determined to be from a non-renal source, the PI will make the decision to proceed with protocol testing and/or randomization.
    * Two out of three consecutive tests greater than or equal to 1+ for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by either a spot urine albumin to creatinine ratio <1000mg/g or a quantitative total urine albumin measurement of < 1g/24 hrs (urine will be screened at admission and repeated if abnormal)
    * Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault <60 mL/min
  * Platelet count below 140,000 K/uL
  * Clinically significant (as determined by the Investigator or Sponsor) abnormalities on laboratory examination that will increase risk to the patient or interfere with data integrity
* Uncontrolled hypothyroidism (abnormal thyroid function tests should be approved by the Investigator)
* History within 6 months of enrollment of screening of drug or alcohol abuse
* History of bleeding diathesis or coagulopathy or clinically significant abnormality in coagulation parameters at enrollment
* Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to enrollment
* Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
* Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated
* Treatment with another investigational drug, biological agent, or device within one month of enrollment, or 5 half-lives of investigational agent, whichever is longer
* Unwilling to comply with contraceptive and lifestyle (diet/exercise) requirements
* Use of any of the following:

  * Use of metreleptin within the last 3 months prior to enrollment
  * Antidiabetic, lipid lowering, or atypical antipsychotic medication, unless on a stable dose for at least 3 months prior to enrollment
  * Insulin unless on a stable daily insulin dose regimen (+/- 20 %) for at least 4 weeks prior to enrollment
  * Use of nicotinic acid or derivatives within the last 4 weeks prior to enrollment
  * Systemic corticosteroids or anabolic steroids within 6 weeks prior to enrollment unless approved by the Investigator
  * Antihypertensive medication unless on a stable dose for at least 4 weeks prior to enrollment
  * Tamoxifen, estrogens or progestins unless on a stable dose for at least 4 months prior to enrollment and dose and regimen expected to remain constant throughout the study
  * Oral anticoagulants unless on a stable dose for at least 4 weeks prior to enrollment and regular clinical monitoring is performed
  * Prior exposure to ISIS 304801
  * Anti-obesity drugs [e.g., the combination of phentermine and extended-release topiramate (Osymia, orlistat (Xenical), liraglutide [rDNA origin] injection (Saxenda) and lorcaserin (Belvig), phentermine, amphetamines, herbal preparations] within 12 weeks prior to screening
  * Any other medication unless stable at least 4 weeks prior to enrollment (occasional or intermittent use of over-the-counter medications will be allowed at Investigator s discretion)
* Blood donation of 50 to 499 mL within 30 days or of >499 mL within 60 days
* Have any other conditions, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-12-23; Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Brown, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared due to the small number of participants

REFERENCES:
- [Background] Jorgensen AB, Frikke-Schmidt R, Nordestgaard BG, Tybjaerg-Hansen A. Loss-of-function mutations in APOC3 and risk of ischemic vascular disease. N Engl J Med. 2014 Jul 3;371(1):32-41. doi: 10.1056/NEJMoa1308027. Epub 2014 Jun 18. PMID 24941082
- [Background] Graham MJ, Lee RG, Bell TA 3rd, Fu W, Mullick AE, Alexander VJ, Singleton W, Viney N, Geary R, Su J, Baker BF, Burkey J, Crooke ST, Crooke RM. Antisense oligonucleotide inhibition of apolipoprotein C-III reduces plasma triglycerides in rodents, nonhuman primates, and humans. Circ Res. 2013 May 24;112(11):1479-90. doi: 10.1161/CIRCRESAHA.111.300367. Epub 2013 Mar 29. PMID 23542898
- [Background] Gaudet D, Alexander VJ, Baker BF, Brisson D, Tremblay K, Singleton W, Geary RS, Hughes SG, Viney NJ, Graham MJ, Crooke RM, Witztum JL, Brunzell JD, Kastelein JJ. Antisense Inhibition of Apolipoprotein C-III in Patients with Hypertriglyceridemia. N Engl J Med. 2015 Jul 30;373(5):438-47. doi: 10.1056/NEJMoa1400283. PMID 26222559
- [Background] Gaudet D, Brisson D, Tremblay K, Alexander VJ, Singleton W, Hughes SG, Geary RS, Baker BF, Graham MJ, Crooke RM, Witztum JL. Targeting APOC3 in the familial chylomicronemia syndrome. N Engl J Med. 2014 Dec 4;371(23):2200-6. doi: 10.1056/NEJMoa1400284. PMID 25470695
- [Derived] Lightbourne M, Startzell M, Bruce KD, Brite B, Muniyappa R, Skarulis M, Shamburek R, Gharib AM, Ouwerkerk R, Walter M, Eckel RH, Brown RJ. Volanesorsen, an antisense oligonucleotide to apolipoprotein C-III, increases lipoprotein lipase activity and lowers triglycerides in partial lipodystrophy. J Clin Lipidol. 2022 Nov-Dec;16(6):850-862. doi: 10.1016/j.jacl.2022.06.011. Epub 2022 Sep 22. PMID 36195542
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-DK-0038.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | ISIS 304801
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ISIS 304801 | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.7 (9.0) | 32.0 (12.7) | 39 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5
Log triglyceride (mg/dL) [Mean (Standard Deviation); unit: log mg/dL] | 2.6 (0.3) | 2.7 (0.0) | 2.6 (0.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Log 10 Fasting Triglycerides.
Description: Change from baseline to 16 weeks in log 10 fasting triglycerides
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: log 10 mg/dl
Arm/Group | Placebo | ISIS 304801
Number analyzed (Participants) | 3 | 2
log 10 mg/dl | 0.1 (0.2) | -0.2 (0.4)

2. Secondary Outcome: Change in Lipolysis Rate (Glycerol)
Description: Change in lipolysis rate measured using stable isotope tracers (Glycerol rate of appearance) (mg/kgLBM/min)
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: mg/kgLBM/min
Arm/Group | Placebo | ISIS 304801
Number analyzed (Participants) | 3 | 2
mg/kgLBM/min | 0.1 (0.6) | 0.3 (2.0)

3. Secondary Outcome: Change in Lipolysis Rate (Palmitate)
Description: Change in lipolysis rate measured using stable isotope tracers (Palmitate rate of appearance) measured in milligrams per kilogram lean body mass per minute (mg/kgLBM/min)
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: mg/kgLBM/min
Arm/Group | Placebo | ISIS 304801
Number analyzed (Participants) | 3 | 2
mg/kgLBM/min | 0.0 (0.1) | -0.2 (0.0)

4. Secondary Outcome: Change From Baseline in Liver Volume
Description: Change from baseline in hepatic steatosis (magnetic resonance spectroscopy) (mL)
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | ISIS 304801
Number analyzed (Participants) | 3 | 2
mL | -114.5 (384.2) | 129.2 (145)

5. Secondary Outcome: Change From Baseline in Hepatic Steatosis
Description: Change from baseline in hepatic steatosis via magnetic resonance spectroscopy
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Placebo | ISIS 304801
Number analyzed (Participants) | 2 | 2
percent | 4.6 (14.9) | -3.8 (0.92)

6. Secondary Outcome: Change in Lipoprotein Lipase Activity
Description: Lipoprotein lipase activity in plasma is measured using blood samples obtained 10 minutes after intravenous infusion of 60 units/kg of unfractionated heparin.
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: nmol FFA/min
Arm/Group | Placebo | ISIS 304801
Number analyzed (Participants) | 3 | 2
nmol FFA/min | -1.6 (1.6) | -3.2 (2.0)

7. Secondary Outcome: Change in Total Body Insulin Sensitivity
Description: Change in total body insulin sensitivity using the hyperinsulinemic euglycemic clamp (mg/kgLBM/min)
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: mg/kgLBM/min
Arm/Group | Placebo | ISIS 304801
Number analyzed (Participants) | 3 | 2
mg/kgLBM/min | -0.1 (2.0) | 0.4 (1.5)

8. Secondary Outcome: Change in HbA1c
Description: Change in hemoglobin A1c (HbA1c) (%)
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Placebo | ISIS 304801
Number analyzed (Participants) | 3 | 2
Percent | 0.6 (0.3) | 0.7 (0.2)

9. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Change in fasting plasma glucose in mg/dL
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | ISIS 304801
Number analyzed (Participants) | 3 | 2
mg/dL | -47 (77) | -71 (100)

10. Secondary Outcome: Plasma ISIS 304801 Level
Description: Measured via a non-compartmental plasma PK analysis of ISIS 304801
Time Frame: 16 weeks
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | ISIS 304801
Number analyzed (Participants) | 3 | 2
ng/mL | 0 (0) | 34.5 (21.5)

ADVERSE EVENTS:
Time Frame: 16 weeks of treatment
Arm/Group | Placebo | ISIS 304801
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/2
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3) | ISIS 304801 (N=2)
Acute Pancreatitis (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3) | ISIS 304801 (N=2)
Injection site reactions (Investigations) | 0 | 2
Elevated liver enzymes (Hepatobiliary disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 1
IV infiltration (Investigations) | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
URI (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/86/NCT02639286/Prot_SAP_000.pdf